CLINICAL TRIAL: NCT00311038
Title: Pilot Study of ONO-1101 in Patients Scheduled for Multi-slice Computed Tomography (CT) Due to Suspected Coronary Artery Disease
Brief Title: Pilot Study of ONO-1101 in Patients Scheduled for Multi-slice CT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONO-1101-24
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Disease
Keywords: ONO-1101; Landiolol Hydrochloride; Multi-slice CT; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — landiolol

INTERVENTIONS:
Drug: ONO-1101

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ONO-1101 in patients scheduled for multi-slice CT.

ELIGIBILITY:
Inclusion Criteria:

1. 20-74 years old
2. Heart rate less than 90 beats/min more than 70 beats/min at entering the CT room

Exclusion Criteria:

1. Previous allergic reactions to contrast agent
2. Renal failure
3. Asthma
4. Other exclusion criteria as specified in the protocol

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-04

PRIMARY OUTCOMES:
heart rate
image quality
safety

CONTACTS AND LOCATIONS:
Overall Officials: Project Leaders Development Planning, Study Director — Ono Pharmaceutical Co. Ltd
Locations (3):
- Japan (3):
  - Hokuriku Region Facility, Hokuriku
  - Kanto Region Facility, Kanto
  - Kyusyu Region Facility, Kyusyu